CLINICAL TRIAL: NCT00922363
Title: An Open Phase I, Dose-escalating, Clinical Trial on the Safety of a New Liposomal Adjuvant System, CAF01, When Given With the Tuberculosis Subunit Vaccine Ag85B-ESAT-6 as Two Injections With Two Months Interval to Healthy Adult Volunteers
Brief Title: Trial on the Safety of a New Liposomal Adjuvant System, CAF01, When Given With the Tuberculosis Subunit Vaccine Ag85B-ESAT-6 as Two Injections With Two Months Interval to Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACAF01-01
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Tuberculosis
Keywords: safety; vaccine; tuberculosis; CAF01; Ag85B-ESAT-6; prevention
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 50 µg Ag85B-ESAT-6 alone (Experimental)
  Interventions: Biological: 50 µg Ag85B-ESAT-6 alone
- 50 µg Ag85B-ESAT-6 + 125/25 µg CAF01 (Experimental)
  Interventions: Biological: 50 µg Ag85B-ESAT-6 + 125/25 µg CAF01
- 50 µg Ag85B-ESAT-6 + 313/63 µg CAF01 (Experimental)
  Interventions: Biological: 50 µg Ag85B-ESAT-6 + 313/63 µg CAF01
- 50 µg Ag85B-ESAT-6 + 625/125 µg CAF01 (Experimental)
  Interventions: Biological: 50 µg Ag85B-ESAT-6 + 625/125 µg CAF01

INTERVENTIONS:
Biological: 50 µg Ag85B-ESAT-6 alone — 0.5 mL solution for injection x 2 (2 months interval)
  Arms: 50 µg Ag85B-ESAT-6 alone
Biological: 50 µg Ag85B-ESAT-6 + 125/25 µg CAF01 — 0,5 mL suspension for injection x 2 (2 months interval)
  Arms: 50 µg Ag85B-ESAT-6 + 125/25 µg CAF01
Biological: 50 µg Ag85B-ESAT-6 + 313/63 µg CAF01 — 0.5 mL suspension for injection x 2 (2 months interval)
  Arms: 50 µg Ag85B-ESAT-6 + 313/63 µg CAF01
Biological: 50 µg Ag85B-ESAT-6 + 625/125 µg CAF01 — 0.5 mL suspension for injection x 2 (2 months interval)
  Arms: 50 µg Ag85B-ESAT-6 + 625/125 µg CAF01

SUMMARY:
The purpose of this study is to evaluate the safety profile of CAF01, administering 50 µg Ag85B-ESAT-6 alone and 50 µg Ag85B-ESAT-6 with three escalating CAF01 dose levels, to four groups of healthy volunteers, injecting two doses with two months interval.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male adult between 18 and 55 years of age
2. Healthy according to medical history and medical examinations at screening
3. Signed informed consent
4. Prepared to grant authorized persons access to medical records
5. Likely to comply with instructions

Exclusion Criteria:

1. History of tuberculosis or known exposure to tuberculosis before (or expected during) the clinical trial
2. Positive Tuberculin Skin Test (TST) result at screening
3. Positive QuantiFERON® -TB Gold In-Tube test result according to the manufacturer's specifications at screening
4. BCG vaccination any time before entering the trial
5. History of or ongoing congenital or acquired immune deficiency, autoimmune disease or thyroid dysfunction
6. Disease affecting the lymphoid organs (Hodgkin's disease, lymphoma, leukaemia, sarcoidosis)
7. ANA-Titer, HBV, HCV, HIV sero-positive at screening
8. C-reactive protein level > 50 mg/L at screening
9. Clinically significant abnormal laboratory test results at screening as assessed by the investigator
10. Severe ongoing viral or bacterial infection that might affect the cell mediated immune response
11. A condition in which repeated blood drawings pose more than minimal risk for the subject, such as haemophilia, other coagulation disorders, or significantly impaired venous access
12. Live vaccine vaccination (MMR, yellow fever, oral typhoid) within 3 months before the first vaccination
13. Immune modulating drugs administration (immunoglobulin, systemic corticosteroids, azathioprine, cyclosporine, infliximab, blood products or vaccines) within 3 months before the first vaccination
14. Known hypersensitivity to any of the vaccine components of the investigational vaccines
15. Intake of another clinical trial product/vaccine within 3 months before the first vaccination or participation in previous clinical trials with the Ag85B-ESAT-6 antigen
16. Pregnant according to a urine pregnancy test at inclusion
17. Females not willing to use contraceptives or breast feeding
18. Has a condition which in the opinion of the investigator is not suitable for participation in the clinical trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Adverse events | one year after first vaccination

SECONDARY OUTCOMES:
Immunogenicity | one year after the first vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Department of infectious diseases, C5-P, LUMC, Leiden, Netherlands